CLINICAL TRIAL: NCT01024777
Title: A Pilot Study to Assess the Relative Safety and Immunology Effects of Low Dose Versus High Dose Cholecalciferol Supplementation in Patients With Multiple Sclerosis
Brief Title: Safety and Immunologic Effect of Low Dose Versus High Dose Vitamin D3 in Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Peter A. Calabresi, Professor of Neurology, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00023005
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Multiple Sclerosis; Vitamin D Deficiency
Keywords: cholecalciferol; multiple sclerosis; vitamin D; D3
MeSH Terms: conditions — Multiple Sclerosis; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- High dose cholecalciferol (Active Comparator): Patients in the high dose arm will receive 10,000 international units of cholecalciferol daily.
  Interventions: Drug: Cholecalciferol
- Low dose cholecalciferol (Active Comparator): Patients enrolled in the low dose arm will receive up to 1000 international units of cholecalciferol daily.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Cholecalciferol (Vitamin D3) 10,000 IU in tablet form will be taken once daily for the duration of the trial (6 months)
  Other Names: Vitamin D3
  Arms: High dose cholecalciferol
Drug: Cholecalciferol — Cholecalciferol (Vitamin D3) 400 IU in tablet form will be taken once daily for the duration of the trial (6 months)
  Other Names: Vitamin D3
  Arms: Low dose cholecalciferol

SUMMARY:
The purpose of this study is to determine the safety and the immunologic effects of supplementation with low-dose and high-dose cholecalciferol (vitamin D3) in patients with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18-55 years (inclusive)
* Serum 25(OH) vitamin D levels between 20-50 ng/mL and a candidate for vitamin D supplementation
* Patients with or without immunomodulatory therapy for RRMS
* Diagnosis of multiple sclerosis

Exclusion Criteria:

* Serum 25(OH) vitamin D deficient level < 20 ng/mL
* High dose vitamin D supplementation in the past 3 months
* Pregnancy
* History of tuberculosis, hyperparathyroidism, sarcoidosis or kidney stones
* Baseline serum creatinine above 1.5
* Hypersensitivity to vitamin D preparations
* Milk allergy
* Unable to consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Assess safety of high dose cholecalciferol in patients with multiple sclerosis | 3-6 months
Assess the effects of cholecalciferol supplementation on serum immune markers in patients with multiple sclerosis | 3-6 months

SECONDARY OUTCOMES:
Assess clinical effects of cholecalciferol supplementation in patients with multiple sclerosis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Calabresi, MD, Principal Investigator — Johns Hopkins University; John Ratchford, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States